CLINICAL TRIAL: NCT04222452
Title: Clinical Consequences of Adults Presenting With hyPophOsphatasia With Special Focus on Gait, Bone micRosTRucture And cognITion: The PORTRAIT Study
Brief Title: The PORTRAIT Study
Acronym: PORTRAIT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: STH20707
Record Dates: First submitted 2019-10-23; First posted 2020-01-10 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-08

CONDITIONS: Hypophosphatasia
Keywords: Burden of disease; Bone microstructure; Cognition; Physical functioning
MeSH Terms: conditions — Hypophosphatasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples (full blood and serum)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypophosphatasia patients (HPP): Patients with known hypophosphatasia (HPP) as diagnosed using genetic testing.
- Controls: Healthy individuals (controls) matched to the cases by gender and age.

SUMMARY:
Clinical Consequences of Adults Presenting with Hypophosphatasia with Special Focus on Gait, Bone Microstructure and Cognition: The PORTRAIT study Hypophosphatasia (HPP) is an inherited condition that leads to weak bones. Early childhood forms are severe and easily recognized. Adult forms can vary in severity. HPP is often missed by doctors or confused with osteoporosis. This is important because the usual osteoporosis treatments may be harmful to patients with HPP and increase the risk of broken bones. One of the reasons it is missed is a lack of research describing the typical features of HPP, so doctors don't recognize the signs, and don't know when or how to test for it. The PORTRAIT Study will help increase understanding of the burden of disease of HPP on patients. The aim is to examine the effects of HPP on bone structure and strength, physical functioning, cognition, and quality of life. Researchers will study adults with HPP and healthy age- and gender-matched individuals. Blood samples will be collected after an overnight fast. Researchers will use these samples to measure markers of HPP and bone health. Medical history and lifestyle, quality of life and cognitive function will be assessed using questionnaires. Bone mineral density, body composition and bone structure and strength will be measured using dual energy x-ray absorptiometry and high resolution peripheral quantitative computed tomography. Physical functioning will be assessed as participants perform a series of physical performance and gait tests. Magnetic resonance images of the lower limbs will be matched-up with the physical functioning data to create patient-specific musculoskeletal models. Cognitive function tests will be performed to assess cognition and mental health. To reveal the burden of disease of HPP, the data collected from patients with HPP will be compared to that collected from healthy controls.

DETAILED DESCRIPTION:
Hypophosphatasia (HPP) is caused by mutations in the tissue non-specific alkaline phosphatase (TNSALP) gene with deficiency in TNSALP activity. This leads to accumulation of inorganic pyrophosphate, a potent inhibitor of bone mineralization, which causes rickets and osteomalacia, and of pyridoxal 5-phosphate (PLP) which causes seizures in neonates but no harm in adults. HPP is also associated with muscle weakness (which is very severe in perinatal and infantile forms) and early tooth loss. The most severe forms of HPP present in infancy, and were fatal until the recent development of TNSALP enzyme replacement therapy, Asfotase Alpha. Adult-onset HPP is less severe. It often presents with fractures of the femur or metatarsals, and so is likely to be misdiagnosed as osteoporosis. Correct diagnosis of HPP is important as the usual osteoporosis treatments, for example bisphosphonates, may be harmful and increase the risk of fracture.

High resolution peripheral quantitative computed tomography (HR-pQCT) is an imaging technique that allows the detailed assessment of BMD, microstructure and strength. HR-pQCT could reveal important information about the effects of HPP on bone microstructural properties.

HPP can also have a significant effect on physical functioning. In infantile HPP, motor function delay is usual but in adult-onset HPP effects on physical functioning are less apparent. These effects can be explored through the use of physical function testing and clinical gait analysis. Cognitive function may be affected by low levels of or inactivity of ALP in the neural tissue (TNALP). Patients with HPP have reported forgetfulness and 'fogginess'.

The aims of the study are to examine the effects of HPP on (i) bone structure and strength, (ii) physical functioning, (iii) cognition and (iv) quality of life (QoL). Researchers will study adults with HPP and healthy individuals. The results will help to determine if there should be a trial of a new drug treatment for adults with HPP. This study forms part of our wider programme of research into HPP.

Researchers will recruit 7 patients with childhood- or adult-presenting HPP (cases), who are known to the Metabolic Bone Clinic at the Metabolic Bone Centre (MBC), Northern General Hospital (NGH), Sheffield. Researchers will also recruit 7 healthy controls matched to the cases by gender and age. Researchers will approach first degree relatives (with their permission) of patients with HPP to offer them genetic testing for HPP. If HPP is confirmed, approach these first degree relatives to invite them to participate in the study, Fasting blood samples will be obtained for measurement of serum or plasma bone alkaline phosphatase (bone ALP), PLP, procollagen type I N-propeptide (PINP), C-terminal telopeptide (CTX) and genetic testing (if not already performed).

Medical history and lifestyle, quality of life and cognitive function will be assessed using questionnaires.

Bone mineral density (BMD) of the lumbar spine, proximal femur and whole body will be measured using dual energy x-ray absorptiometry (DXA). Whole body composition will also be determined by DXA. Trabecular and cortical BMD and bone microstructure and strength will be examining using HR-pQCT of the distal radius and tibia.

Physical functioning will also be assessed. Participants will undergo a series of physical performance tests/gait analysis tests. Chair rises (sit to stand), a timed up and go test. A 10 m walking test and a 4 stair climb will be used to assess muscle strength. A modified performance oriented mobility assessment-gait (MPOMA-G) will also be performed. Recordings of the kinematics, ground reaction forces, electromyography (EMG) data and muscle function will be made using a motion capture system. This will allow the quantification of joint kinematics and kinetics and of muscular pattern activation during the execution of a number of different motor skills. Lower limb magnetic resonance imaging (MRI), with the participants dressed in a set of MRI visible markers, will allow the registration of the MRI and physical functioning/gait data enhancing the participant's specific musculoskeletal modelling.

Cognitive function tests (a Montreal Cognitive Assessment) will be performed to assess the burden of disease of HPP on cognitive and mental health as forgetfulness and 'fogginess' have been reported by patients.

The results from the various assessments performed will be compared between the age-gender matched cases and controls using paired samples t-tests. For each test, the mean difference, 95% confidence interval and associated p-value will be reported. In the event of the normality assumption of the paired samples t-test being violated comparisons will be made using the non-parametric Wilcoxon signed rank test. The burden of disease of HPP on bone quality (i.e. BMD, bone structure and strength), mental health, cognition, QoL, pain, physical functioning and gait will be examined using Spearman Rank Correlation.

ELIGIBILITY:
Inclusion Criteria:

HPP PATIENTS (CASES)

* Clinical diagnosis of HPP (with or without previous genetic test confirmation)
* Evidence of burden of disease (HPP) including abnormal gait, muscle weakness, pain, recurring fractures, slow healing fractures and/or bone deformities
* Age ≥ 18 years
* Able and willing to participate in the study
* Able to give written informed consent

HEALTHY INDIVIDUALS (CONTROLS)

* Healthy men and women with normal bone mineral density (defined as a DXA bone mineral density T- score at the lumbar spine or total hip greater than -1).
* Age ≥ 18 years
* Able and willing to participate in the study
* Able to give written informed consent

Exclusion Criteria:

HPP PATIENTS (CASES)

* Individuals with BMI<18, or BMI>30 kg/m2
* Other conditions known to affect serum ALP and PLP
* Coeliac disease, B12 deficiency, untreated hypothyroidism, Wilson's disease
* Taking nutritional supplements containing vitamin B6 within past two weeks
* History of, or current:

Severe ischaemic heart disease, rheumatoid arthritis, ankylosing spondylitis, cancer (concurrent)

* History of, or current neurological diseases affecting the neuromuscular system including Parkinson's disease, CVA, muscular dystrophy, myasthenia, cerebral trauma, peripheral neuropathy
* Treatment for more than 3 months in a year or under treatment with oral corticosteroids
* History of any long term immobilization (duration greater than three months)
* Conditions or surgery which prevent the acquisition or analysis of musculoskeletal images
* Use of medications or treatment known to affect bone metabolism other than calcium/vitamin D supplementation.
* Alcohol intake greater than 21 units per week
* Pregnant or breast feeding

HEALTHY INDIVIDUALS (CONTROLS)

* Individuals with BMI<18, or BMI>30 kg/m2
* Other conditions known to affect serum ALP and PLP
* Coeliac disease, B12 deficiency, untreated hypothyroidism, Wilson's disease
* Taking nutritional supplements containing vitamin B6 within the past two weeks
* Bilateral fractures of the distal radius and/or distal tibia
* History of, or current conditions known to affect bone metabolism and bone mineral density including diagnosed skeletal disease or arthritis, chronic hepatic or renal disease, Coeliac and/or other malabsorption syndromes, hyperparathyroidism, hyperthyroidism and/or diagnosed endocrine disorders, hypocalcaemia or hypercalcemia, diagnosed restrictive eating disorder, diabetes mellitus
* History of, or current severe ischaemic heart disease, rheumatoid arthritis, ankylosing spondylitis, cancer (concurrent)
* History of, or current neurological diseases affecting the neuromuscular system including Parkinson's disease, CVA, muscular dystrophy, myopathies, myasthenia, cerebral trauma, peripheral neuropathy
* Treatment for more than 3 months in a year or under treatment with oral corticosteroids
* History of any long term immobilization (duration greater than three months)
* Conditions or surgery which prevent the acquisition or analysis of musculoskeletal images
* Use of medications or treatment known to affect bone metabolism other than calcium/vitamin D supplementation.
* Alcohol intake greater than 21 units per week
* Conditions that currently impact on gait
* Pregnant or breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with HPP (cases) and healthy individuals (controls)
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Clinical consequences and disease burden of HPP on the total score (balance + Gait) achieved during the Tinetti Performance Oriented Mobility Assessment (POMA) | Through study completion, average 18 months
  Differences in gait: HPP patients versus healthy controls

SECONDARY OUTCOMES:
Clinical consequences and disease burden of HPP on volumetric Bone Mineral Density (vBMD, in g/cm3) | Through study completion, average 18 months
  Differences in bone microstructure: HPP patients versus healthy controls
Clinical consequences and disease burden of HPP on the total score achieved during the Montreal Cognitive Assessment (MoCA) Test | Through study completion, average 18 months
  Differences in cognitive function: HPP patients versus healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Richard Eastell, MD, Principal Investigator — University of Sheffield
Locations (1):
- The University of Sheffield, Sheffield, South Yorkshire, United Kingdom